CLINICAL TRIAL: NCT03094689
Title: Cold Water Immersion in the Recovery of Clinical, Biochemical, Functional and Neuromuscular Markers of Muscle Damage of 10km Street Runners: Clinical, Randomized and Blinded Trial
Brief Title: Cold Water Immersion in the Recovery of Markers of Muscle Damage of 10km Street Runners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Wouber Hérickson de Brito Vieira, Principal Investigator, Clinical Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.441.252
Record Dates: First submitted 2017-01-05; First posted 2017-03-29 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Health Behavior
Keywords: Physical activity; Muscle pain; Cryotherapy
MeSH Terms: conditions — Health Behavior; Motor Activity; Myalgia

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Control group (No Intervention)
- Immersion group (Experimental): They will be immersed in a barrel of 200 liters of water (without ice) at room temperature, according to local conditions of temperature and humidity (Natal county - RN). They will be immersed to the height of the iliac crests for 10 minutes.
  Interventions: Other: Water immersion
- Cold water immersion group (Experimental): They will be immersed in a barrel of 200 liters of ice water at an average temperature of 10 ° C for 10 minutes. They will be immersed to the height of the iliac crests.
  Interventions: Other: Cold water immersion

INTERVENTIONS:
Other: Cold water immersion
  Arms: Cold water immersion group
Other: Water immersion
  Arms: Immersion group

SUMMARY:
Objective: To analyze the effect of cold water immersion (CWI) on the recovery of clinical, biochemical, functional and neuromuscular markers of muscle damage in 10 km street runners.

Materials and Methods: This is a randomized, blinded trial in which 30 subjects, 10 km street runners, were randomly divided into three groups: control (gC), immersion (gI) and CWI (gCWI). The runners will be evaluated for clinical (subjective perception of exertion), biochemical (serum CK), functional (unipodal triple hop distance and shuttle test time) and neuromuscular variables by means of isokinetic variables (peak torque, total work and fatigue index). Volunteers will perform pre-assessment, immediately post-race and post-intervention, and 24-hour post-intervention. The data will be expressed by mean and standard deviation, analyzed in the statistical package SPSS 20.0. A significance level of 5% and a 95% confidence interval will be considered for all measures.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 30 kg/m2;
* Street runners for at least 6 months;
* Week frequency of at least 3 times;
* Do not present cardiopathies, muscles and neurological diseases;

Exclusion Criteria:

* Hypersensitivity or allergies to cryotherapy;
* Unable to complete the 10 km event on the day of the evaluation;
* Do not complete or perform any of the study procedures for any reason (phobias, do not withstand the exposure time).

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Subjective perception of pain. | Up to 10 weeks
  The subjective perception of pain will be measured by means of the visual analogic scale based on the self-report of the level of pain.